CLINICAL TRIAL: NCT01031992
Title: Efficacy of Tranexamic Acid Taken Orally in Patients With Hereditary Hemorrhagic Telangiectasia
Brief Title: Tranexamic Acid and Epistaxis in Hereditary Hemorrhagic Telangiectasia (HHT)
Acronym: TAHHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Collaborators: Pharmacia GmbH, Erlangen, Germany (Unknown); Baxter Healthcare Corporation (Industry)
Responsible Party: Universitätskliniken des Saarlandes
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAHHT; 141CHC9008-001 (Other: BfArM (German Federal Institute for Drugs and Medical Products))
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
Keywords: Hereditary hemorrhagic telangiectasia; Rendu-Osler-Weber syndrome; Epistaxis; Nosebleeds; Anemia; Tranexamic acid; Antifibrinolytics
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis; Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Experimental): First verum (3 times 1 g Tranexamic acid daily) for three months, than placebo for 3 months.
  Interventions: Drug: Tranexamic acid first, than placebo
- Group II (Experimental): First placebo for 3 months, than verum for 3 months (3 times 1 g Tranexamic acid daily).
  Interventions: Drug: First placebo, than Tranexamic acid.

INTERVENTIONS:
Drug: Tranexamic acid first, than placebo — For 3 months Tranexamic acid 3 times daily 1 g taken orally, followed by placebo for 3 months.
  Arms: Group I
Drug: First placebo, than Tranexamic acid. — First placebo for 3 months, than tranexamic acid 3 times daily 1 g for 3 months.
  Arms: Group II

SUMMARY:
Hereditary hemorrhagic telangiectasia (HHT, Rendu-Osler-Weber Syndrome) is associated with frequent nosebleeds in the majority of cases. Several reports in the literature support the use of antifibrinolytics like Tranexamic acid to reduce nosebleeds. The objectives of the study are to test if Tranexamic acid taken orally can

1. improve anemia (lead to an increased hemoglobin level)
2. reduce nosebleeds.

ELIGIBILITY:
Inclusion Criteria:

* hereditary hemorrhagic telangiectasia with nosebleeds and desire to be treated.

Exclusion Criteria:

* pregnant,
* minor,
* had an increased risk of thrombotic events (history or signs of cerebrovascular events, cardiac arrhythmias, biochemically increased coagulation parameters),
* renal insufficiency,
* a history of massive hematuria or defects of color vision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2002-03; Primary Completion 2002-08 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Change of hemoglobin level within the phases. | Beginning and end of each 3 months period.

SECONDARY OUTCOMES:
Mean epistaxis score (daily duration multiplied by mean subjective daily intensity) | Measured once a day during each 3 months period

CONTACTS AND LOCATIONS:
Overall Officials: Urban W Geisthoff, Priv.-Doz. Dr.med., Principal Investigator — Medical Faculty of the University of the Saarland and Hospitals of the City of Cologne
Locations (1):
- Universitätskliniken des Saarlandes, HNO-Abteilung, Homburg, Saarland, Germany

REFERENCES:
- [Derived] Geisthoff UW, Seyfert UT, Kubler M, Bieg B, Plinkert PK, Konig J. Treatment of epistaxis in hereditary hemorrhagic telangiectasia with tranexamic acid - a double-blind placebo-controlled cross-over phase IIIB study. Thromb Res. 2014 Sep;134(3):565-71. doi: 10.1016/j.thromres.2014.06.012. Epub 2014 Jun 16. PMID 25005464